CLINICAL TRIAL: NCT02261701
Title: Rehabilitation After Rotator Cuff Repair a Randomised Controlled Study
Brief Title: Rehabilitation After Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LTV-426521; ACJCKFVästerås (Other: UppsalaU)
Record Dates: First submitted 2014-09-03; First posted 2014-10-10 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Rotator Cuff Injury
Keywords: shoulder surgery; rotator cuff injury; rehabilitation; function; pain; quality of life
MeSH Terms: conditions — Rotator Cuff Injuries; Pain | interventions — Early Ambulation; Postoperative Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early mobilization (Experimental): Intervention is early mobilization, four weeks immobilization postsurgery with collar´n cuff only.
  Interventions: Other: Early mobilization
- Post surgery shoulder lock (Other): Post surgery shoulder lock with abduction cushion 3 weeks and after this period collar´n cuff 3 weeks
  Interventions: Other: Post surgery shoulder lock

INTERVENTIONS:
Other: Early mobilization — Early mobilization, collar´n cuff 4 weeks post surgery and after this light exercises start and no further bandage.
  Other Names: Collar´n cuff 4 weeks post surgery and early mobilization
  Arms: Early mobilization
Other: Post surgery shoulder lock — Post surgery: Shoulder lock with abduction cushion, additionally 3 weeks with collar´n cuff, and after this period light exercises are allowed and nu further bandage.
  Other Names: Shoulder lock three weeks post surgery
  Arms: Post surgery shoulder lock

SUMMARY:
A new postoperative regimen with a new bandage technique after surgery results in a better shoulder function and quality of life after surgery - than traditional postoperative regimen with shoulder lock and abductor cushion.

DETAILED DESCRIPTION:
A new postoperative regimen , with a new bandage technique with shorter immobilization time and without shoulder lock, is supposed to results in a better shoulder function 6 and 12 months after surgery. Function is measured by Constant score, pain with VAS and quality of life with EQ5D, 3 and 12 months after surgery. The two treatment groups are compared.

ELIGIBILITY:
Inclusion Criteria:

* planned shoulder surgery, rotator cuff repair

Exclusion Criteria:

* not swedish speaking
* reoperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Shoulder function | 6 months after surgery
  Shoulder function is assessed by Constant score

SECONDARY OUTCOMES:
Pain | 6 months after surgery
  Visual analogue scale

OTHER OUTCOMES:
EQ-5D | 6 months after surgery
  Quality of life
Quality of life shoulder specific | 6 months after surgery
  Western Ontario Rotator Cuff Index (WORC)
Pain | 12 months after surgery
  Visual analogue scale
Euro quality of Life 5D | 12 months after surgery
  Quality of life
Quality of life shoulder specific | 12 months after surgery
  Western Ontario Rotator Cuff Index (WORC)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Christin Johansson, PhD, Study Chair — Center for Clinical Research County Västmanland, Sweden
Locations (1):
- Department of Orthopaedic surgery, Physiotherapy, Västerås, Västmanland County, Sweden

IPD SHARING:
Plan to Share IPD: No